CLINICAL TRIAL: NCT01632813
Title: Neurocognitive Development in Children With Congenital Heart Disease: Growing Into Deficit
Brief Title: Leuven Growing Into Deficit Follow-up Study
Acronym: Leuven-GID
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Greet Van den Berghe, Head of Dept Intensive Care Medicine, KU Leuven
Other Study IDs: Leuven-GID
Record Dates: First submitted 2012-06-29; First posted 2012-07-03 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Heart Defects, Congenital; Critical Illness; Mental Processes; Child
Keywords: neurocognitive testing; critical illness; executive function; intelligence
MeSH Terms: conditions — Heart Defects, Congenital; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CHD group: Seven-year-old children with CHD who were four years old when they participated in Paediatric ICU follow-up study (i.e. first follow-up time point) (Neurocognitive development of children four years after critical illness and treatment with tight glucose control, Clinical Trials # NCT00214916). The children of the CHD-group underwent cardiac surgery as infants (=<1year).
- Control group: Seven-year-old healthy control children who were four years old when they participated in Paediatric ICU follow-up study (i.e. first follow-up time point) (Neurocognitive development of children four years after critical illness and treatment with tight glucose control, Clinical Trials # NCT00214916). These children have never undergone cardiac surgery.

SUMMARY:
The key objective of the Leuven growing-into-deficit (GID) follow-up-study is to test the hypothesis that children with a congenital heart disease (CHD) show more neurocognitive impairment at the second follow-up at 7 years old than at the first follow-up at the age of 4, compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Seven-year-old children with CHD and healthy control children who were four years old when they participated in Paediatric ICU follow-up study (i.e. first follow-up time point) (Neurocognitive development of children four years after critical illness and treatment with tight glucose control, Clinical Trials # NCT00214916). The children of the CHD-group underwent cardiac surgery as infants (=<1year).

Exclusion Criteria:

* Genetic syndromes (Down, 22q11del), known to result in neurocognitive impairment
* IQ < 70
* Lack of baseline neurocognitive measurements during first follow-up
* Date of birth before February 2005

Ages: 84 Months to 89 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Seven-year-old children with CHD and healthy seven-year-old control children
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
reaction time (RT) and error rates of inhibitory control (Response Organization Objects, ROO) (Amsterdam Neuropsychological Tasks, ANT) | one testpoint at age of 7 years

SECONDARY OUTCOMES:
reaction time (RT) and error rates of cognitive flexibility (ROO, ANT) and working memory (Memory Search - Objects 2 Keys, ANT) | one testpoint at age of 7 years
Mean RT + standard deviation (SD) of RT on computerized alertness task (Baseline Speed, ANT) | one testpoint at age of 7 years
Number of taps on computerized tapping tasks (ANT) | one testpoint at age of 7 years
IQ measures (Revised Wechsler Preschool and Primary Scale of Intelligence, WPPSI-R) | one testpoint at age of 7 years
Visual-Motor Integration total standard score (VMI) | one testpoint at age of 7 years
Child Behavior CheckList T-scores for internalizing and externalizing problems | one testpoint at age of 7 years
Pediatric Quality of Life Inventory - Generic Score Scales (PedsQL) to quantify quality of life | one testpoint at age of 7 years
Behavior Rating Inventory of Executive Function (BRIEF) to measure executive functions (parent and teacher version) | one testpoint at age of 7 years
Teacher Report Form (TRF) T-scores for internalizing and externalizing problems at school | one testpoint at age of 7 years
Incidence of medical problems (e.g. head trauma), interventions and operations since first follow-up | one testpoint at age of 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Mesotten, MD PhD, Principal Investigator — KU Leuven
Locations (1):
- Dept Intensive Care Medicine, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- [Background] Vlasselaers D, Milants I, Desmet L, Wouters PJ, Vanhorebeek I, van den Heuvel I, Mesotten D, Casaer MP, Meyfroidt G, Ingels C, Muller J, Van Cromphaut S, Schetz M, Van den Berghe G. Intensive insulin therapy for patients in paediatric intensive care: a prospective, randomised controlled study. Lancet. 2009 Feb 14;373(9663):547-56. doi: 10.1016/S0140-6736(09)60044-1. Epub 2009 Jan 26. PMID 19176240
- [Derived] Sterken C, Lemiere J, Van den Berghe G, Mesotten D. Neurocognitive Development After Pediatric Heart Surgery. Pediatrics. 2016 Jun;137(6):e20154675. doi: 10.1542/peds.2015-4675. PMID 27245833